CLINICAL TRIAL: NCT07144969
Title: Comparison of the Effect of Chewing Gum and Honey on Postoperative Recovery and Complications in Ileostomy Reversal
Brief Title: Chewing Gum vs Honey in Postoperative Recovery After Ileostomy Reversal: A Study Comparing Their Effects on Bowel Function, Complications, and Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Hospital Lahore (Other)
Responsible Party: Principal Investigator, Shahroze Wajid, Dr. Shahroze Wajid, Mayo Hospital Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IleostomyReversalHoneyvsGum
Record Dates: First submitted 2025-07-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Ileostomy Closure; Gum Chewing; Honey; Postoperative Recovery; Postoperative Complications After Gastrointestinal Operations
Keywords: ileostomy; reversal; stoma; closure; honey; gum; recovery; complications; ERAS; pilot; randomized control trial
MeSH Terms: interventions — Honey; Chewing Gum

STUDY DESIGN:
Intervention Model Description: This was a prospective, single-blinded, parallel-group randomized controlled pilot trial with a 1:1 allocation ratio conducted at Mayo Hospital, Lahore. Thirty patients undergoing ileostomy reversal were randomized into two groups using a lottery method: Group A received chewing gum, and Group B received natural honey, both starting 24 hours postoperatively. Group A chewed gum for 5 minutes every 4 hours, while Group B consumed half a tablespoon of honey every 4 hours. Primary outcomes (time to pass flatus, stools and bowel sounds) and secondary outcomes (time to full feeds, Postoperative ileus, Intraabdominal infection, Nausea and vomiting, Postoperative hospital stay) were recorded every 8 hours.
Masking Description: Selection bias were addressed by randomly assigning the participants to the groups. Performance bias cannot be eliminated due to different surgeons performing the ileostomy reversal surgery. Detection bias were addressed by keeping the participants unaware of what group they are assigned to and because of the objective nature of the outcome variables. There was still some detection bias in some respects involving the subjective opinion of the participants e.g. pain score. Intention-to-treat analysis were done to address attrition bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Intervention: Chewing gum every 4 hours (Experimental)
  Interventions: Dietary Supplement: gum chewing
- Group B - Intervention: Natural honey every 4 hours (Active Comparator)
  Interventions: Dietary Supplement: Honey

INTERVENTIONS:
Dietary Supplement: Honey — Group B patients were asked to eat one half tablespoon of natural honey every 4 hours
  Arms: Group B - Intervention: Natural honey every 4 hours
Dietary Supplement: gum chewing — Group A patients were asked to chew gum for 5 minutes every 4 hours
  Arms: Group A - Intervention: Chewing gum every 4 hours

SUMMARY:
Title: Comparison of the effect of chewing gum and honey on postoperative recovery and complications in ileostomy reversal - a pilot randomized controlled trial Background: Ileostomy reversal is associated with postoperative complications such as ileus, delayed gastrointestinal function recovery (GIFR), and infections. Chewing gum (sham feeding) and honey have been proposed as cost-effective interventions to enhance recovery, but their comparative efficacy remains underexplored.

Objective: To evaluate the effects of chewing gum versus honey on postoperative recovery and complications in patients undergoing ileostomy reversal.

Methods: A prospective single-blinded pilot randomized controlled trial is to be conducted at Mayo Hospital, Lahore, involving 30 patients (15 per group). Group A received chewing gum, while Group B received honey, starting 24 hours postoperatively. Primary outcomes included time to bowel sounds, flatus, and feces. Secondary outcomes were time to full feeds, intraabdominal infections, postoperative ileus, nausea/vomiting, and length of hospital stay. Data significance was set at p < 0.05.

DETAILED DESCRIPTION:
"Comparison of the Effect of Chewing Gum and Honey on Postoperative Recovery and Complications in Ileostomy Reversal - A Pilot Randomized Controlled Trial"

1. Introduction

   Background

   Ileostomy reversal is a standard procedure following temporary diversion surgeries, yet it's frequently complicated by issues such as ileus, delayed gastrointestinal function recovery (GIFR), infections, and longer hospital stays. Enhanced Recovery After Surgery (ERAS) protocols have emphasized early feeding and noninvasive stimulatory interventions like sham feeding (e.g., chewing gum), aiming to improve outcomes by accelerating return of bowel function. Honey, long known for its medicinal and antimicrobial properties, has also shown promise in enhancing gastrointestinal health and wound healing. However, its use postoperatively in gastrointestinal surgery, particularly ileostomy reversal, has not been well studied.

   Rationale

   This study addresses the research gap concerning the comparative effects of chewing gum and honey in enhancing postoperative recovery following ileostomy reversal. It aims to evaluate their efficacy in improving outcomes and reducing complications, using a pilot randomized controlled trial design.
2. Objective

   To compare the effects of chewing gum and honey on:

   Time to bowel sounds, flatus, feces Time to full feeds Postoperative ileus Intraabdominal infection Nausea and vomiting Postoperative hospital stay
3. Methods

Study Design

A prospective, single-blinded pilot randomized controlled trial was conducted at the West Surgical Ward, Mayo Hospital Lahore.

Participants

Sample size: 30 patients (15 per group) Inclusion: Adults (>18 years) undergoing ileostomy reversal after >1 month of stoma creation Exclusion: Malignancy, Irritable bowel disease (IBD), inability to chew/swallow, preexisting complications

Interventions

Group A (Gum): Chewed gum for 5 minutes every 4 hours, starting 24 hours postop Group B (Honey): Consumed ½ tablespoon honey every 4 hours, starting 24 hours postop

Outcomes

Primary: Time to bowel sounds, flatus, feces Secondary: Time to full feeds, PONV, pain score, discharge time, hospital stay, complications

Randomization & Blinding

Randomization was done using a lottery method. The study was single-blinded: participants were unaware of which group they were assigned to.

Data Collection

Standardized protocols for auscultation, patient self-reporting, and case report documentation were used. All participants completed the trial without loss to follow up.

ELIGIBILITY:
Inclusion Criteria:

* All patients of age more than 18 years with an Ileostomy
* Undergoing surgery involving reversal of an Ileostomy i.e., Loop Ileostomy, Double Barrel Ileostomy, Ileocolostomy or End Ileostomy
* Time from fashioning of ileostomy to its reversal is of a duration greater than 1 month

Exclusion Criteria:

* Patients with existing complications as mentioned above in the operative definition of postoperative complications
* Patients with malignancy
* Patients with inflammatory bowel disease
* Patients who cannot communicate well
* Patients who have difficulty chewing or swallowing
* Patients who are prohibited from oral intake by the surgeon
* Patients having undergone Ileostomy reversal more than 1 day before being included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Time to pass flatus | Assessed by asking the patient if they have passed flatus every 8 hours starting from 24 hours after the ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  Defined as the time, in hours, between the completion of surgery and the documented passage of the first objectively confirmed flatus by auscultation or direct observation
Time to bowel sounds | Assessed by ausculating the patients' abdomen to listen to the presence or absence of bowel sounds every 8 hours starting from 24 hours after the ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  Defined as the time, in hours, between the completion of surgical closure and the first audible auscultation of non-continuous, high-pitched bowel sounds originating from the reconnected intestine, documented by a trained healthcare professional using a stethoscope placed over the lower quadrants of the abdomen
Time to pass feces | Assessed by asking the patient if they have passed stool every 8 hours starting from 24 hours after the Ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  Defined as the time, in hours, between the completion of surgery and the documented first independent bowel movement, excluding any stool manually evacuated or stimulated by laxatives

SECONDARY OUTCOMES:
Time to full feeds | Assessed by asking the patient if they have taken full feeds every 8 hours starting from 24 hours after the ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  Defined as the time, in hours, between the surgery and the first point at which the patient tolerates and consumes a regular, unrestricted diet without experiencing any significant postoperative gastrointestinal complications (e.g., nausea, vomiting, abdominal pain, ileus) for a predetermined timeframe (i.e., 24 hours)
Postoperative Pain | Assessed by asking the patient about their abdominal pain using a Visual Analog score from 0 to 10 every 8 hours starting from 24 hours after the ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  Postoperative pain in stoma reversal surgery was defined as the subjective pain intensity experienced by the patient at rest or during movement, assessed using the Visual Analog Scale (VAS). The VAS consists of a 10 cm horizontal line anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10), with patients marking the point on the line that best represented their pain intensity.
Postoperative nausea and vomiting (PONV) | Assessed by asking the patient about the number of vomiting episodes or nausea they had every 8 hours starting from 24 hours after the ileostomy reversal procedure up to 5 days (144 hours) postoperatively.
  PONV was defined as the number of episodes of documented postoperative nausea/emesis or administration of a rescue antiemetic
Length of postoperative stay/ Time to discharge | Assessed by calculating the time of hospital stay (in hours) between the Ileostomy reversal surgery up to 5 days (144 hours) postoperatively.
  Defined as the time, in hours, of the postoperative hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Shahroze Wajid, Postgraduate Resident Surgery, Principal Investigator — West Surgical Ward, Mayo Hospital, Lahore
Locations (1):
- Mayo Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
In light of patient doctor confidentiality, the individual patient data will not be disclosed

REFERENCES:
- [Background] Behera BK, Misra S, Tripathy BB. Systematic review and meta-analysis of safety and efficacy of early enteral nutrition as an isolated component of Enhanced Recovery After Surgery [ERAS] in children after bowel anastomosis surgery. J Pediatr Surg. 2022 Aug;57(8):1473-1479. doi: 10.1016/j.jpedsurg.2021.07.020. Epub 2021 Jul 28. PMID 34417055
- [Background] Gil-Vargas M, Saavedra-Pacheco MS, Coral-Garcia MA. Early Feeding versus Traditional Feeding in Children with Ileostomy Closure. J Indian Assoc Pediatr Surg. 2022 Mar-Apr;27(2):223-226. doi: 10.4103/jiaps.JIAPS_388_20. Epub 2022 Mar 1. PMID 35937106
- [Background] Peng Y, Xiao D, Xiao S, Yang L, Shi H, He Q, Xu H, Zhu X, Zhong W, Yu J. Early enteral feeding versus traditional feeding in neonatal congenital gastrointestinal malformation undergoing intestinal anastomosis: A randomized multicenter controlled trial of an enhanced recovery after surgery (ERAS) component. J Pediatr Surg. 2021 Sep;56(9):1479-1484. doi: 10.1016/j.jpedsurg.2021.02.067. Epub 2021 Mar 18. PMID 33838898
- [Background] Hsu YC, Szu SY. Effects of Gum Chewing on Recovery From Postoperative Ileus: A Randomized Clinical Trail. J Nurs Res. 2022 Oct 1;30(5):e233. doi: 10.1097/jnr.0000000000000510. PMID 35951432
- [Background] Park SH, Choi MS. Meta-Analysis of the Effect of Gum Chewing After Gynecologic Surgery. J Obstet Gynecol Neonatal Nurs. 2018 May;47(3):362-370. doi: 10.1016/j.jogn.2018.01.011. Epub 2018 Mar 3. PMID 29505755
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Bhatti S, Malik YJ, Changazi SH, Rahman UA, Malik AA, Butt UI, Umar M, Farooka MW, Ayyaz M. Role of Chewing Gum in Reducing Postoperative Ileus after Reversal of Ileostomy: A Randomized Controlled Trial. World J Surg. 2021 Apr;45(4):1066-1070. doi: 10.1007/s00268-020-05897-1. Epub 2021 Jan 5. PMID 33403448
- [Background] Lin Z, Li Y, Wu J, Zheng H, Yang C. Nomogram for prediction of prolonged postoperative ileus after colorectal resection. BMC Cancer. 2022 Dec 6;22(1):1273. doi: 10.1186/s12885-022-10377-x. PMID 36474177
- [Background] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Background] Atkins CS, Tubog TD, Schaffer SK. Chewing Gum After Radical Cystectomy With Urinary Diversion for Recovery of Intestinal Function: A Systematic Review and Meta-Analysis. J Perianesth Nurs. 2022 Aug;37(4):467-473. doi: 10.1016/j.jopan.2021.10.003. Epub 2022 Mar 8. PMID 35272926
- [Background] Luo J, Xia M, Zhang C. The Effects of Chewing Gum on Reducing Anxiety and Stress: A Meta-Analysis of Randomized Controlled Trials. J Healthc Eng. 2022 Jan 31;2022:8606693. doi: 10.1155/2022/8606693. eCollection 2022. PMID 35140905
- [Background] de Gaay Fortman DPE, Kroon HM, Bedrikovetski S, Fitzsimmons TR, Dudi-Venkata NN, Sammour T. A snapshot of intraoperative conditions to predict prolonged postoperative ileus after colorectal surgery. ANZ J Surg. 2022 Sep;92(9):2199-2206. doi: 10.1111/ans.17784. Epub 2022 May 17. PMID 35579059
- [Background] Li K, Wang D, Zhang X, Yang J, Chen X. Efficacy of early enteral nutrition versus total parenteral nutrition for patients with gastric cancer complicated with diabetes mellitus: A systematic review and meta-analysis. Nutr Diet. 2022 Feb;79(1):129-139. doi: 10.1111/1747-0080.12721. PMID 35233912
- [Background] Akbulut S, Dogan Z, Baskiran A, Elbe H, Turkoz Y. Effect of a honey and arginine-glutamine-hydroxymethylbutyrate mixture on the healing of colon anastomosis in rats immunosuppressed with tacrolimus. Biotech Histochem. 2019 Oct;94(7):514-521. doi: 10.1080/10520295.2019.1601257. Epub 2019 Apr 15. PMID 30983411
- [Background] Negahi AR, Hosseinpour P, Vaziri M, Vaseghi H, Darvish P, Bouzari B, Mousavie SH. Comparison of Honey versus Polylactide Anti-Adhesion Barrier on Peritoneal Adhesion and Healing of Colon Anastomosis in Rabbits. Open Access Maced J Med Sci. 2019 May 25;7(10):1597-1601. doi: 10.3889/oamjms.2019.284. eCollection 2019 May 31. PMID 31210807
- [Background] Khan A, Haris M, Rehman M, Khan MJ, Abdullah, Haris S. Early Postoperative Complications and Surgical Anatomy After Ileostomy Reversal Among the Population of Khyber Pakhtunkhwa, Pakistan. Cureus. 2021 Nov 17;13(11):e19660. doi: 10.7759/cureus.19660. eCollection 2021 Nov. PMID 34958658
- [Background] Venara A, Neunlist M, Slim K, Barbieux J, Colas PA, Hamy A, Meurette G. Postoperative ileus: Pathophysiology, incidence, and prevention. J Visc Surg. 2016 Dec;153(6):439-446. doi: 10.1016/j.jviscsurg.2016.08.010. Epub 2016 Sep 23. PMID 27666979
- [Background] Aktas A, Kayaalp C, Ates M, Dirican A. Risk factors for postoperative ileus following loop ileostomy closure. Turk J Surg. 2020 Dec 29;36(4):333-339. doi: 10.47717/turkjsurg.2020.4911. eCollection 2020 Dec. PMID 33778391
- [Background] Eroglu O, Deniz T, Kisa U, Comu FM, Kaygusuz S, Kocak OM. The effect of different types of honey on healing infected wounds. J Wound Care. 2018 Oct 1;27(Sup10):S18-S25. doi: 10.12968/jowc.2018.27.Sup10.S18. PMID 30307813
- [Background] Suresh K, Thomas SV, Suresh G. Design, data analysis and sampling techniques for clinical research. Ann Indian Acad Neurol. 2011 Oct;14(4):287-90. doi: 10.4103/0972-2327.91951. PMID 22346019
- [Background] Tashkandi H. Honey in wound healing: An updated review. Open Life Sci. 2021 Oct 6;16(1):1091-1100. doi: 10.1515/biol-2021-0084. eCollection 2021. PMID 34708153
- [Background] Chapman SJ, Thorpe G, Vallance AE, Harji DP, Lee MJ, Fearnhead NS; Association of Coloproctology of Great Britain and Ireland Gastrointestinal Recovery Group. Systematic review of definitions and outcome measures for return of bowel function after gastrointestinal surgery. BJS Open. 2018 Oct 1;3(1):1-10. doi: 10.1002/bjs5.102. eCollection 2019 Feb. PMID 30734010
- [Background] Eteraf-Oskouei T, Najafi M. Traditional and modern uses of natural honey in human diseases: a review. Iran J Basic Med Sci. 2013 Jun;16(6):731-42. PMID 23997898
- [Background] Scepankova H, Combarros-Fuertes P, Fresno JM, Tornadijo ME, Dias MS, Pinto CA, Saraiva JA, Estevinho LM. Role of Honey in Advanced Wound Care. Molecules. 2021 Aug 7;26(16):4784. doi: 10.3390/molecules26164784. PMID 34443372
- [Background] Saikaly SK, Khachemoune A. Honey and Wound Healing: An Update. Am J Clin Dermatol. 2017 Apr;18(2):237-251. doi: 10.1007/s40257-016-0247-8. PMID 28063093
- [Background] Bode CO, Ademuyiwa AO, Elebute OA. Formal saline versus honey as escharotic in the conservative management of major omphaloceles. Niger Postgrad Med J. 2018 Jan-Mar;25(1):48-51. doi: 10.4103/npmj.npmj_159_17. PMID 29676346
- [Background] Canzan F, Caliaro A, Cavada ML, Mezzalira E, Paiella S, Ambrosi E. The effect of early oral postoperative feeding on the recovery of intestinal motility after gastrointestinal surgery: Protocol for a systematic review and meta-analysis. PLoS One. 2022 Aug 18;17(8):e0273085. doi: 10.1371/journal.pone.0273085. eCollection 2022. PMID 35980900
- [Background] Grass F, Pache B, Butti F, Sola J, Hahnloser D, Demartines N, Hubner M. Stringent fluid management might help to prevent postoperative ileus after loop ileostomy closure. Langenbecks Arch Surg. 2019 Feb;404(1):39-43. doi: 10.1007/s00423-018-1744-4. Epub 2019 Jan 3. PMID 30607532
- [Background] Daams F, Wu Z, Lahaye MJ, Jeekel J, Lange JF. Prediction and diagnosis of colorectal anastomotic leakage: A systematic review of literature. World J Gastrointest Surg. 2014 Feb 27;6(2):14-26. doi: 10.4240/wjgs.v6.i2.14. PMID 24600507
- [Background] Ng ZQ, Levitt M, Platell C. The feasibility and safety of early ileostomy reversal: a systematic review and meta-analysis. ANZ J Surg. 2020 Sep;90(9):1580-1587. doi: 10.1111/ans.16079. Epub 2020 Jun 28. PMID 32597018
- [Background] Peltrini R, Magno G, Pacella D, Iacone B, Rizzuto A, Bracale U, Corcione F. Postoperative Morbidity Following Loop Ileostomy Reversal after Primary Elective or Urgent Surgery: A Retrospective Study with 145 Patients. J Clin Med. 2023 Jan 5;12(2):452. doi: 10.3390/jcm12020452. PMID 36675381
- [Background] Ghosh A, Biswas SK, Basu KS, Biswas SK. Early Feeding after Colorectal Surgery in Children: Is it Safe? J Indian Assoc Pediatr Surg. 2020 Sep-Oct;25(5):291-296. doi: 10.4103/jiaps.JIAPS_132_19. Epub 2020 Sep 1. PMID 33343110
- [Background] Aznan MI, Khan OH, Unar AO, Tuan Sharif SE, Khan AH, Syed Abd Aziz SH, Zakaria AD. Effect of Tualang honey on the anastomotic wound healing in large bowel anastomosis in rats-A randomized controlled trial. BMC Complement Altern Med. 2016 Jan 23;16:28. doi: 10.1186/s12906-016-1003-6. PMID 26803744
- [Background] Fernandez-Galvez A, Rivera S, Duran Ventura MDC, de la Osa RMR. Nutritional and Educational Intervention to Recover a Healthy Eating Pattern Reducing Clinical Ileostomy-Related Complications. Nutrients. 2022 Aug 20;14(16):3431. doi: 10.3390/nu14163431. PMID 36014936
- [Background] Rahimi VB, Shirazinia R, Fereydouni N, Zamani P, Darroudi S, Sahebkar AH, Askari VR. Comparison of honey and dextrose solution on post-operative peritoneal adhesion in rat model. Biomed Pharmacother. 2017 Aug;92:849-855. doi: 10.1016/j.biopha.2017.05.114. Epub 2017 Jun 10. PMID 28618654
- [Background] Amanollahi O, Azizi B. The comparative study of the outcomes of early and late oral feeding in intestinal anastomosis surgeries in children. Afr J Paediatr Surg. 2013 Apr-Jun;10(2):74-7. doi: 10.4103/0189-6725.115025. PMID 23860050
- [Background] Chu L, Wang H, Qiu S, Shao B, Huang J, Qin Q, He Y, Xue J, Li X, Huang X, Huang R. Risk Factors of Delayed Recovery of Gastrointestinal Function After Ileostomy Reversal for Rectal Cancer Patients. Cancer Manag Res. 2021 Jun 29;13:5127-5133. doi: 10.2147/CMAR.S311715. eCollection 2021. PMID 34234556
- [Background] Madan S, Sureshkumar S, Anandhi A, Gurushankari B, Keerthi AR, Palanivel C, Kundra P, Kate V. Comparison of Enhanced Recovery After Surgery (ERAS) Pathway Versus Standard Care in Patients Undergoing Elective Stoma Reversal Surgery- A Randomized Controlled Trial. J Gastrointest Surg. 2023 Nov;27(11):2667-2675. doi: 10.1007/s11605-023-05803-9. Epub 2023 Aug 24. PMID 37620661
- [Background] Westfall KM, Rivard SJ, Suwanabol PA, Albright JJ, Ramm CA, Cleary RK. Postoperative Oral Rehydration and Regimented Follow-up Decrease Readmissions After Colorectal Surgery That Includes Ileostomies. Dis Colon Rectum. 2024 Feb 1;67(2):313-321. doi: 10.1097/DCR.0000000000002935. Epub 2023 Sep 12. PMID 37703205
- [Background] Ahmed MR, Sayed Ahmed WA, Khamess RE, Youwakim MS, El-Nahas KM. Efficacy of three different regimens in recovery of bowel function following elective cesarean section: a randomized trial. J Perinat Med. 2018 Sep 25;46(7):786-790. doi: 10.1515/jpm-2017-0389. No abstract available. PMID 29451863
- [Background] Patel S, Duncan A. Anaesthesia and intestinal anastomosis. BJA Educ. 2021 Nov;21(11):433-443. doi: 10.1016/j.bjae.2021.06.001. Epub 2021 Sep 21. No abstract available. PMID 34707889
- [Background] Scott MJ, Baldini G, Fearon KC, Feldheiser A, Feldman LS, Gan TJ, Ljungqvist O, Lobo DN, Rockall TA, Schricker T, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 1: pathophysiological considerations. Acta Anaesthesiol Scand. 2015 Nov;59(10):1212-31. doi: 10.1111/aas.12601. Epub 2015 Sep 8. PMID 26346577
- [Background] Baraza W, Wild J, Barber W, Brown S. Postoperative management after loop ileostomy closure: are we keeping patients in hospital too long? Ann R Coll Surg Engl. 2010 Jan;92(1):51-5. doi: 10.1308/003588410X12518836439209. PMID 20056062
- [Background] Girard E, Messager M, Sauvanet A, Benoist S, Piessen G, Mabrut JY, Mariette C. Anastomotic leakage after gastrointestinal surgery: diagnosis and management. J Visc Surg. 2014 Dec;151(6):441-50. doi: 10.1016/j.jviscsurg.2014.10.004. Epub 2014 Oct 22. PMID 25455960
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT07144969/Prot_SAP_ICF_000.pdf